CLINICAL TRIAL: NCT06244927
Title: Replantation Following Complete Penile Amputation: Summary of Perioperative Experience and Treatment Strategies Before and After Case Study
Brief Title: Replantation Following Complete Penile Amputation
Status: Completed | Type: Observational
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0699
Record Dates: First submitted 2024-01-19; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Penile Amputation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Only 20 patients undergo replantation following penile amputation were investigate, only 1group: Patients undergo surgery.
  Interventions: Procedure: Replantation surgery

INTERVENTIONS:
Procedure: Replantation surgery — Surgery

SUMMARY:
The goal of this observational study Replantation following Complete Penile Amputation a case series before and after study is to help andrologist and urologists deal with such rare male emergencies easily in emergency situation. There are only limited case reports of penile amputation, a rare urological emergency with a low treatment success rate, and there are still no advanced, detailed surgical or perioperative treatment plans.The main question[s] it aims to answer are:

•The investigators used questionnaire to ask participants who undergo replantation surgery to reply. These are the International Index of Erectile Function (IIEF) before and after surgery; the International Prostate Symptom Score (IPSS) estimate for urination after surgery; the Quality of Life index (QoL) estimate, which characterized quality of life into 7 categories: happy (0), satisfied (1), general satisfied (2), not bad (3), not too satisfied (4), distressed (5), and terrible (6). The appearance satisfaction score was based on four levels: from unsatisfactory (1), slight unsatisfactory (2), satisfactory (3) to very satisfactory(4).

Participants (Patients) only need to reply question above. This is observational before and after case study.

DETAILED DESCRIPTION:
Twenty participants (aged 6-58 years) who were treated at investigators' hospital over the past years and ultimately underwent surgery and follow-up assessment were included. The relevant research was approved by the Ethics Committee of Sir Run Run Shaw Hospital, Approval NO.: 2023-0699. All 20 amputated phalli were adequately preserved; the neurovascular structures in the proximal stump were readily identified and in a suitable condition for anastomosis. All of these parameters were evaluated by the investigators, who believed that anastomosis could be attempted. The surgery was performed under the guidance of the investigators, and the same surgical methods were used. Surgical methods and perioperative processes were performed as described below. The participants' preoperative erectile functions and urination scores are shown in Table 1. Each of the participants and their families desired penis replantation after the accident, even if the amputation occurred because of a psychological disorder. A participant may not be willing to undergo replantation due to psychological issues, but their families are supportive of replantation. And surgeons believe that there is high probability of successful anastomosis creation. This participant was constraint to undergoing treatment. The participants' details can be found in Table 1. The investigators used the International Index of Erectile Function (IIEF) before and after surgery; the International Prostate Symptom Score (IPSS) estimate for urination after surgery; the Quality of Life index (QoL) estimate, which characterized quality of life into 7 categories: happy (0), satisfied (1), general satisfied (2), not bad (3), not too satisfied (4), distressed (5), and terrible (6). The appearance satisfaction score was based on four levels: from unsatisfactory (1), slight unsatisfactory (2), satisfactory (3) to very satisfactory(4)

ELIGIBILITY:
Inclusion Criteria:

Patients who received replantation surgeries following penile amputation. And complete follow-up data.

Exclusion Criteria:

Patients who not received replantation surgeries following penile amputation. Or Incomplete follow-up data.

Ages: 6 Years to 58 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who received replantation surgeries following penile amputation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
International Index of Erectile Function (IIEF) | 6 months
  Revealing the quality of the patient's erectile function

SECONDARY OUTCOMES:
International Prostate Symptom Score (IPSS) | 6 months
  Revealing the quality of the patient's urination

CONTACTS AND LOCATIONS:
Overall Officials: Hanchao Liu, Study Chair — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data can be shared upon reasonable request